CLINICAL TRIAL: NCT00725881
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase 1/2 Dose-Range-Finding Study to Evaluate the Safety, Efficacy and PK of Multiple Once Daily Intravenous Doses of TSC in Patients With Intermittent Claudication
Brief Title: Safety, Efficacy, and Pharmacokinetics (PK) Study of Trans Sodium Crocetinate (TSC) in Patients With Intermittent Claudication
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diffusion Pharmaceuticals Inc (Industry)
Responsible Party: Kim M. Whitten, PharmD, RAC, Diffusion Pharmaceuticals LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DP100-301
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Intermittent Claudication
Keywords: PAD; Peripheral arterial disease; Peripheral artery disease; Intermittent claudication; IC; atherosclerosis; leg pain; walking pain
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease; Atherosclerosis | interventions — trans-sodium crocetinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 1 (Experimental): .25 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 2 (Experimental): .5 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 3 (Experimental): .75 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 4 (Experimental): 1.0 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 5 (Experimental): 1.25 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 6 (Experimental): 1.5 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 7 (Experimental): 1.75 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 8 (Experimental): 2.0 mg/kg TSC
  Interventions: Drug: Trans sodium crocetinate (TSC)
- 9 (Placebo Comparator): 5.0 mL 0.9% normal saline
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: Trans sodium crocetinate (TSC) — Once-daily bolus intravenous injections in a superficial vein of the arm via syringe over a period of up to 2 minutes. Each patient will receive up to 5 doses given on 5 consecutive days
  Arms: 1; 2; 3; 4; 5; 6; 7; 8
Drug: 0.9% normal saline — A total volume of 5.0 mL normal saline will be dosed in a superficial vein of the arm via syringe over a period of up to 2 minutes.
  Arms: 9

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of multiple, once-daily, intravenous doses of trans sodium crocetinate (TSC). The effectiveness of TSC in alleviating the symptoms of intermittent claudication (IC) will also be assessed.

DETAILED DESCRIPTION:
Peripheral Artery Disease (PAD) is a manifestation of systemic atherosclerosis, and patients with PAD commonly manifest symptoms of intermittent claudication (IC) such as cramping, aching, or fatigue in the calf muscles provoked by activity. In PAD, arterial occlusions lead to decreased leg blood flow during exercise or walking and the pain associated with this ischemia is IC. The diffusion of oxygen from blood to muscle could be a component of the overall decreased delivery or deficit of oxygen (hypoxia) to skeletal muscle resulting in symptoms in PAD patients. The overall goal of the development of TSC as a treatment for PAD is to allow for enhanced diffusion of oxygen through the plasma to alleviate the symptoms caused by the hypoxia in the tissues.

This double-blinded, placebo-controlled clinical trial will randomize up to 48 patients at up to 8 clinical research sites in the US. In addition to safety and pharmacokinetic assessments conducted during the trial, the primary endpoint of the study will be demonstrated from standardized, graded exercise treadmill tests conducted throughout the study. The clearly measurable parameters will be peak walking time (PWT) and claudication onset time (COT) comparing baseline and after TSC or placebo and are well-established endpoints accepted by the medical community and regulatory authorities for IC clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 or older, male or female
* 6-mo. history of walking limitation or symptoms of intermittent claudication (IC) in at least 1 lower limb, severity of which has not changed in the past 3 mo. and diagnosed by principal investigator as clinically stable Fontaine Stage II peripheral artery disease (PAD)
* Diagnosis of PAD secondary to atherosclerosis
* If ankle-brachial index (ABI) is > 1.3 or cannot be measured in either leg, vascular etiology documented by toe-brachial index (TBI) ≤ 0.7 in at least 1 leg
* Claudication severity, meds. for the treatment of coronary artery disease (CAD), PAD and IC, and exercise habits should be clinically stable for 3 mo. prior to Screening (SCRN) and during study. Pt. is not likely to change smoking and/or exercise habits during study
* On an exercise treadmill test (ETT), peak walking time (PWT) of at least 1 min., but no more than 12 min. at Baseline
* Willing and able to discontinue Pletal or Trental for 21 days before SCRN and during study
* Antihypertensive therapy, cholesterol-lowering therapy, chronic oral nitrates, and diabetic therapy have been stable for 30 days prior to SCRN
* Willing and able to provide written, signed, informed consent after the nature of the study has been explained and prior to any research-related procedures
* Willing and able to comply with all study-related procedures
* Sexually active patients must use an acceptable method of contraception while participating in the study
* Females of childbearing potential must have a negative pregnancy test at SCRN and have additional pregnancy tests during the study

Exclusion Criteria:

* Pregnant or lactating
* Current or history of critical limb ischemia (CLI)
* Pts. in whom artery insufficiency in the lower extremity is the result of acute limb ischemia (ALI) or an immunological or inflammatory non-atherosclerotic disorder
* Pts. in whom walking impairment due to pain is the result of other non-atherosclerotic co-morbid conditions
* A surgical intervention to alleviate symptoms of IC or PAD-specific endovascular intervention or cardiovascular surgery within 3 mo. of SCRN
* Walking limited by reasons other than claudication
* Conditions other than IC of significant severity that could confound PWT on the ETT
* Concurrent severe congestive heart failure (CHF)
* Life-threatening ventricular arrhythmias, unstable angina, and/or myocardial infarction (MI) within 3 mo. before enrollment (ENRL)
* Coronary artery bypass grafting or percutaneous coronary intervention within 4 mo. before ENRL
* Renal and/or carotid revascularization procedure within 3 mo. of ENRL
* Transient ischemic attack (TIA) within 3 mo. before ENRL
* Deep vein thrombosis (DVT) within 3 mo. before ENRL
* Severe chronic obstructive pulmonary disease (COPD)
* Thrombocytopenia
* Undergoing hemodialysis or peritoneal dialysis
* Pts. w/immunocompromised conditions, organ transplant recipients and/or need for immunosuppressive therapy
* Neurological dementia
* Stroke
* Clinically significant electrocardiogram (ECG) change during or after ETT at SCRN or Baseline visit(s)
* Cerebrovascular infarct within 3 mo. of SCRN
* Poorly controlled type 1 or type 2 diabetes at SCRN
* History of migraine headaches within last 12 mo.
* Patients with clinically significant abnormal hematology labs or blood chemistry labs
* Body mass index > 35
* Hypertension at SCRN defined as resting BP values of > 170 mmHg systolic and/or > 110 mmHg diastolic
* Hypotension at SCRN defined as resting BP values < 100 mmHg systolic or < 55 mmHg diastolic or symptomatic hypotension
* Previous treatment with any formulation of TSC
* Known allergy or hypersensitivity to any excipient (gamma-cyclodextrin, mannitol, glycine) of TSC formulation
* Previous treatment with gene therapy or other VEGF-related treatment within 12 mo. of SCRN
* Patients with recent history of alcoholism or drug abuse, or severe emotional, behavioral, or psychiatric problems
* Patients receiving experimental medications or participating in other study using an experimental drug or procedure within 45 days prior to ENRL

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety (laboratory tests, vital signs, ECG, physical exam, pulse oximetry) and pharmacokinetic assessments | Screening, Baseline, Dose 1, Dose 2, Dose 3, Dose 4, Dose 5, 5-Day Follow-up, 14-Day Follow-up

SECONDARY OUTCOMES:
Change in peak walking time (PWT) and claudication onset time (COT) in an exercise treadmill test | Baseline, Dose 1, Dose 5, 5-Day Follow-up

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cardiology, P.C., Birmingham, Alabama
  - Radiant Research, Inc., Santa Rosa, California
  - Stanford University School of Medicine, Division of Cardiovascular Medicine, Stanford, California
  - Andrews Research and Education, Pensacola, Florida
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Trials of Texas, Inc., San Antonio, Texas

REFERENCES:
- [Derived] Mohler ER 3rd, Gainer JL, Whitten K, Eraso LH, Thanaporn PK, Bauer T. Evaluation of trans sodium crocetinate on safety and exercise performance in patients with peripheral artery disease and intermittent claudication. Vasc Med. 2011 Oct;16(5):346-53. doi: 10.1177/1358863X11422742. PMID 22003000